CLINICAL TRIAL: NCT05610774
Title: Using Optic Nerve Sheath Diameter to Monitor Intracranial Tension in Pre-Eclamptic Parturient Receiving Magnesium Sulfate in Combination With Dexmedetomidine
Brief Title: Optic Nerve Sheath Diameter in Pre-Eclamptic Parturient Receiving Magnesium Sulfate Combined With Dexmedetomidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, lecturer of anesthesia and surgical ICU, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC 23.9.2022
Record Dates: First submitted 2022-11-01; First posted 2022-11-09 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Preeclampsia Severe; Optic Nerve Sheath Diameter
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (D) (Experimental): Patients will receive a loading dose of iv dexmedetomidine followed by a maintenance infusion.
  Interventions: Drug: Dexmedetomidine
- Group (C) (Placebo Comparator): patients will receive saline loading and infusion
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — pre-eclamptic Patients will receive a loading dose of iv dexmedetomidine (0.5 ug/kg) diluted in 50 ml saline and given over 10 min, followed by a maintenance infusion of (0.2 ug/kg/h) diluted in 200 ml saline till The sedation scores on the Richmond Agitation and Sedation Scale was -2 to +1 (lightly sedated to restless).
  Arms: Group (D)
Drug: Saline — pre-eclamptic patients will receive 50 ml saline loading for 10 min followed by 200 ml saline infusion
  Arms: Group (C)

SUMMARY:
Dexmedetomidine was reported to effectively reduce cerebral metabolism and ICP by decreasing cerebrospinal fluid pressure in patients with cerebral tumors or head injuries that require craniotomy. However, it was also reported to exhibit no effect on ICP. the effect of MgSO4 associated with dexmedetomidine on ONSD in severely pre-eclamptic parturient has been understudied . Though this study aims to evaluate the effect of dexmedetomidine infusion on raised ICP in severely pre-eclamptic parturients using ocular ultrasonography to determine ONSD as a measure of ICP.

DETAILED DESCRIPTION:
Dexmedetomidine, a highly selective α-2-receptor agonist, is a first-line sedative medication in ICU and has been increasingly used for obstetric anesthesia. Dexmedetomidine, which provides light sedation, possesses analgesic, sympatholytic, anxiolytic properties and attenuates the stress response without significant respiratory depression. In addition, dexmedetomidine-induced stimulation of postsynaptic alpha-2 adrenergic receptor on the cerebral blood vessels can cause cerebral vasoconstriction and decrease cerebral blood flow. However, the effects of dexmedetomidine on ICP are controversial.

Clinical signs of raised ICP are not specific and often difficult to interpret, especially during pregnancy and pre-eclampsia. Though the use of invasive devices is considered a gold standard in the measurement of ICP, Ocular sonography is a promising bedside tool, which serves as a noninvasive, readily available, and cost-effective means for indirectly measuring ICP.

Bedside ultrasound can be used as a point-of-care tool for rapidly measuring the optic nerve sheath diameter (ONSD), which is a validated indirect means for measuring ICP. An increase in ICP reflects as a raised ONSD since the optic nerve is surrounded by Dural sheath and cerebrospinal fluid (CSF) containing subarachnoid space, which is distensible in the retrobulbar segment, particularly when CSF pressures rise.

ELIGIBILITY:
Inclusion Criteria:

* aged18 to 40 years with
* at least 36 weeks gestation
* admitted with diagnosis of severe pre-eclampsia and scheduled to receive Magnesium Sulphate therapy before delivery

Exclusion Criteria:

* Presence of ocular wound or Prior ocular surgery
* emergency cases, and evidence of fetal compromise
* HELLP syndrome (hemolysis, elevated liver enzymes, and low platelet levels)
* Chronic hypertension
* Hyperthyroidism, and diabetes mellitus
* Presence of pre-existing chronic lung and/or cardiac diseases
* Presence of pre-existing chronic renal and/or hepatic diseases
* Presence of any chronic diseases of central nervous system.
* known allergies to the tested drug.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter (ONSD) measurments following Drug administration | Baseline (before starting MgSO4 therapy) then at 1, 6, 12 and 24 hours postoperative

SECONDARY OUTCOMES:
The incidence of raised ICP in severe pre-eclampsia | Baseline (before starting MgSO4 therapy), and during 24 hours postoperative.
  ONSD >5.0 mm
Sedation Score | every 2 hours after drug infusion, till 24 postoperative hours
  the Richmond Agitation and Sedation Scale (RASS), on which scores range from -5 [unresponsive] to +4 [combative].
Heart Rate (HR) | Baseline (before starting MgSO4 therapy) then every 2 hours till 24 postoperative hours
mean arterial pressure (MAP) changes. | Baseline (before starting MgSO4 therapy) then every 2 hours till 24 postoperative hours
The duration of hospital stay | one month after delivery
  defined as time from the day of operation to the day of discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Rafik Amin, Banhā, Qalyubia Governorate, Egypt